CLINICAL TRIAL: NCT01596348
Title: Perceived Exercise Benefits, Barriers and Preferences Among Swiss Rheumatoid Arthritis Patients
Brief Title: Exercise Perceptions and Preferences Among Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Collaborators: University of Lausanne Hospitals (Other)
Other Study IDs: PR_Ex
Record Dates: First submitted 2011-06-21; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Exercise; Barriers; Benefits; Preferences; Stages of change
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients: Patients with Rheumatoid Arthritis

SUMMARY:
The purpose of the study is to analyse exercise behaviour of rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis
* Age 30 to 80 years

Exclusion Criteria:

* Language difficulties and no help from family members or friends

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected in the Rheumatology Department of the Centre Hospitalier universitaire Vaudois in Lausanne.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Exercise status
  * Trained
  * Active
  * Irregularly active
  * Partially active
  * Inactive
Exercise stages of change
  Prochaska 1992:
  * Precontemplation
  * Contemplation
  * Preparation
  * Action
  * Maintenance
Perceived exercise benefits
  Questionnaire developped by YH based on existing qualitive studies
Perceived exercise barriers
  Questionnaire developped by Brittain et al. 2011
Exercise preferences
  Developped by YH based on previous studies

SECONDARY OUTCOMES:
Functional status
  Health Assessment Questionanire (Guillemin et al. 1991)
Pain
  Visual analogue scale (VAS)
Fatigue
  VAS
Disease activity
  Disease activity score 28 (DAS 28), based on the number of tender and swollen joints and the erythrocite sedimentation rate (ESR)
Quality of life
  Arthritis Impact Measurement Scales 2

CONTACTS AND LOCATIONS:
Overall Officials: Alexander KL So, PhD, FRCP, Study Director — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Département de l'Appareil Locomoteur, Lausanne, Switzerland